CLINICAL TRIAL: NCT05832164
Title: Prevalence of Frailty in Individuals With HIV Infection and Age Older Than 60 Years, Factors Associated and 6-month Effectiveness of a Multifactorial Intervention: HIDRA360
Brief Title: Effectiveness of a Multifactorial Intervention in Frailty Individuals With HIV Infection: HIDRA360
Acronym: HIDRA360
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Costa del Sol (Other)
Responsible Party: Principal Investigator, Julian Olalla Sierra, Medical Specialist, Department of Internal Medicine, Hospital Costa del Sol, Marbella (Malaga,) Spain, Hospital Costa del Sol
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0368-N-22
Record Dates: First submitted 2023-04-12; First posted 2023-04-27 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Frailty Syndrome; HIV Infections
Keywords: Dependence; Nutrition; Physical activity; Polymedication;
MeSH Terms: conditions — Frailty; HIV Infections; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study design consists of two stages: a descriptive cross-sectional study to assess the prevalence of frailty in a cohort of HIV patients and, subsequently, a quasi-experimental before/after study without equivalent control group to evaluate the effectiveness of a multifactorial intervention. The intervention will be offered to all patients, regardless of their frailty, pre-frailty or robustness status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multifactorial intervention (Experimental): HIV patients
  Interventions: Other: Multifactorial intervention

INTERVENTIONS:
Other: Multifactorial intervention — * Adherence to a Mediterranean diet.
  * Progressive aerobic and anaerobic exercise program.
  * Review of polypharmacy
  * Group socialization activities

SUMMARY:
The goal of this quasi-experimental before/after study without equivalent control group is to to describe the prevalence of frail, pre-fragile and robust individuals in the study group before and after a multifactorial intervention in in frail HIV patients.

The main questions it aims to answer are after a multifactorial intervention:

1. To describe the sociodemographic, viroimmunological and ART exposure factors of fragile individuals compared to pre-fragile and robust individuals.
2. To describe adherence to the Mediterranean diet in frail individuals compared to pre-frail and robust individuals.
3. To describe the presence of anxiety and depression in frail individuals with respect to pre-fragile and robust individuals.
4. To describe the analytical parameters and inflammatory markers of frail individuals with respect to pre-fragile and robust individuals.
5. To describe the diversity and composition of the intestinal microbiota of frail individuals with respect to pre-fragile and robust individuals.
6. To describe the body composition of frail individuals with respect to pre-fragile and robust individuals.
7. To describe the factors associated with progression to frailty or robustness after six months of a multifactorial intervention.

DETAILED DESCRIPTION:
After the baseline visit, a multifactorial intervention will be carried out consisting of:

* Distribution of short videos (10-15', in a number not exceeding 10), focused on the maintenance of a Mediterranean and balanced diet, developed by the nutrition service of our hospital. If the pandemic situation allows it, explanatory sessions will be organized with the same purpose of physical presence.
* Distribution of short videos (10-15', in a number not exceeding 10) focused on the implementation and adherence to a progressive program of aerobic and anaerobic exercise, developed by the physiotherapy service of our hospital. If the pandemic situation allows it, explanatory sessions will be organized for the same purpose of physical presence.
* Review of polypharmacy by the HIV Unit of our hospital.
* Communication with the NGO Avance Positivo for the development of group socialization activities.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection of at least 6 months' duration after initial diagnosis
* Ability to sign the informed consent form
* Stable residence in our health area

Exclusion Criteria:

* Barthel Index<90
* Prognosis of less than one year of life at the discretion of the investigator.
* Inability to complete the study (8 months) as judged by the investigator or the patient
* Presence of Child stage C cirrhosis, end-stage renal failure (Fge by CKD-EPI<10 mL/min or dialysis in any form), dementia.
* Bone fracture within the last 3 months that interferes with gait or prehensile strength in the judgement of the investigator.
* Diagnosis prior to inclusion in the study of diseases requiring the use of chemotherapy, radiotherapy or non-minor surgery.
* End of chemotherapy or radiotherapy in the three months prior to study entry
* Major surgery in the three months prior to study entry
* Current diagnosis of wasting syndrome
* Active neoplasm at the time of study entry, except for non-melanoma skin cancer or anal carcinoma in situ

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Determine change in frailty status after multifactorial intervention | 6 months
  To assess change in frailty status: frail, pre-frail and robust; in cohort of patients before and after multifactorial intervention. It will be assessed through Fried's Phenotype which includes 5 classic criteria: slowed gait speed, poor physical activity, self-reported physical tiredness, unintentional weight loss and muscle weakness. With three or more criteria the patient will be considered as frail, 1 or 2 as pre-frail and robust in absence.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Costa del Sol, Marbella, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No